CLINICAL TRIAL: NCT00975884
Title: Safety and Immunogenicity Study of GSK Biologicals' Influenza Vaccine GSK2340272A in Adults Aged 18 Years and Above
Brief Title: Study to Evaluate Immunogenicity & Safety of an Investigational Influenza Vaccine in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113630; 2009-015008-25 (EudraCT Number)
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-02

CONDITIONS: Influenza
Keywords: GSK Bio's influenza vaccine GSK2340272A; influenza infection; Influenza vaccine
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- GSK2340272A (D21) GROUP (Experimental): Healthy male or female adults, above 18 years of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21 (D21).
  Interventions: Biological: GSK investigational vaccine GSK2340272A
- GSK2340272A (M6) GROUP (Experimental): Healthy male or female adults, above 18 years of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Month 6 (M6).
  Interventions: Biological: GSK investigational vaccine GSK2340272A

INTERVENTIONS:
Biological: GSK investigational vaccine GSK2340272A — Two intramuscular injections

SUMMARY:
The objective of this study is to evaluate the immunogenicity and safety of GSK Biologicals' investigational vaccine GSK2340272A.

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged 18 years or above at the time of the first vaccination.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Satisfactory baseline medical assessment by history and physical examination. Stable health status is defined as the absence of a health event satisfying the definition of a serious adverse event, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within one month prior to enrolment.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination, and
* has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period. Potential subjects in the follow-up phase of a prior investigational study may be enrolled if the investigator's judgment is that it will have no effect on safety, reactogenicity, or immunogenicity endpoints in this study, and that it does not violate the protocol requirements of the prior trial.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of an axillary temperature >= 37.5ºC, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination. NOTE: The subject may be vaccinated at a later date, provided symptoms have resolved, vaccination occurs within the window specified by the protocol, and all other eligibility criteria continue to be satisfied.
* Diagnosed with cancer, or treatment for cancer, within the past 3 years.
* Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
* Persons with a history of histological-confirmed basal cell carcinoma of the skin successfully treated with local excision only are excepted and may enrol within 3 years of diagnosis, but other histological types of skin cancer require a 3 year untreated and disease-free window as above.
* Women who are disease-free 3 years or more after treatment for breast cancer and receiving long-term prophylactic hormonal therapy are excepted and may enrol.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Chronic administration of immunosuppressants or other immune modifying drugs within 6 months of study enrolment or planned administration during the study period.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrolment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome.
* Clinically or virologically confirmed influenza infection within 6 months preceding the study start.
* Administration of any vaccines within 30 days before vaccination.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Pregnant or lactating female
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any conditions which, in the opinion of the investigator, prevents the subjects from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2009-09-14 (Actual); Primary Completion 2010-04-30 (Actual); Study Completion 2010-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- France (4):
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Poitiers

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Duval X, Caplanusi A, Laurichesse H, Deplanque D, Loulergue P, Vaman T, Launay O, Gillard P. Flexibility of interval between vaccinations with AS03A-adjuvanted influenza A (H1N1) 2009 vaccine in adults aged 18-60 and >60 years: a randomized trial. BMC Infect Dis. 2012 Jul 23;12:162. doi: 10.1186/1471-2334-12-162. PMID 22824474
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113630 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113630 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113630 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113630 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113630 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113630 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 313 subjects enrolled in the study, 7 subjects did not receive any vaccination.
Groups:
- GSK2340272A (D21) GROUP: Healthy male or female adults, divided into subjects between and including 18 to 60 years of age and subjects older than 60 years of age (>60), who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21 (D21).
- GSK2340272A (M6) GROUP: Healthy male or female adults, divided into subjects between and including 18 to 60 years of age and subjects older than 60 years of age (>60), who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Month 6 (M6).
Period: Overall Study
Arm/Group | GSK2340272A (D21) GROUP | GSK2340272A (M6) GROUP
Started | 184 | 122
Completed | 168 | 107
Not Completed | 16 | 15
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 9 | 9
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340272A (D21) GROUP | GSK2340272A (M6) GROUP | Total
Number analyzed (Participants) | 184 | 122 | 306
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.8 (16.8) | 51.6 (16.0) | 52.3 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 63 | 155
  Male | 92 | 59 | 151
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African Heritage / African American | 4 | 2 | 6
  Geographic ancestry: Asian - Central/South Asian Heritage | 0 | 1 | 1
  Geographic ancestry: Asian - East Asian Heritage | 3 | 1 | 4
  Geographic ancestry: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Geographic ancestry: White - Arabic / North African Heritage | 3 | 3 | 6
  Geographic ancestry: White - Caucasian / European Heritage | 174 | 114 | 288

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted (SCR) Subjects for Haemagglutination Inhibition (HI) Antibodies
Description: Seroconversion was defined as: For initially seronegative subjects [antibody titer below (<) 1:10 post to vaccination], antibody titer greater than or equal to (≥) 1:40 after vaccination; For initially seropositive subjects (antibody titer ≥ 1:10 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was A/California/7/2009 (H1N1)v-like influenza (Flu A/CAL/7/09). The Committee for Medicinal Products for Human Use (CHMP) criterion was fulfilled if the point estimate for SCR was > 40% in subjects 18 to 60 years of age or > 30% for subjects above 60 years of age.
Time Frame: At Day 21
Population: The According-To-Protocol (ATP) cohort for immunogenicity at Day 21 included all eligible subjects, for whom 1 dose of study vaccine was administered and assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 days after the first vaccine dose.
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340272A 18-60 YEARS SUB-GROUP: Pooled group for healthy male or female adults, between and including 18 to 60 years of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21 and at Month 6.
- GSK2340272A > 60 YEARS SUB-GROUP: Pooled group for healthy male or female adults, older than 60 years of age (>60), who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21 and at Month 6.
Arm/Group | GSK2340272A 18-60 YEARS SUB-GROUP | GSK2340272A > 60 YEARS SUB-GROUP
Number analyzed (Participants) | 160 | 136
Participants | 154 | 121

2. Primary Outcome: Number of Subjects Who Were Seroprotected (SPR) for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40, that usually is accepted as indicating protection. The CHMP criterion was fulfilled if the post-vaccination point estimate for SPR was > 70% in subjects 18 to 60 of age or > 60% for subjects above 60 years of age.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 YEARS SUB-GROUP | GSK2340272A > 60 YEARS SUB-GROUP
Number analyzed (Participants) | 160 | 136
Participants | 156 | 125

3. Primary Outcome: Percentage of Seroconverted (SCR) Subjects for HI Antibodies
Description: as for outcome 1
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | GSK2340272A 18-60 YEARS SUB-GROUP | GSK2340272A > 60 YEARS SUB-GROUP
Number analyzed (Participants) | 160 | 136
Percentage of subjects | 96.3 [92.0 to 98.6] | 89.0 [82.5 to 93.7]

4. Primary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: GMFR, also called seroconversion factor (SCF), was defined as the fold increase in serum HI geometric mean titers (GMTs) post-vaccination compared to pre-vaccination. The flu strain assessed was Flu A/CAL/7/09. The criterion was fulfilled if the point estimate for GMFR was > 2.5 in subjects 18 to 60 years of age or > 2 for subjects above 60 years of age.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2340272A 18-60 YEARS SUB-GROUP | GSK2340272A > 60 YEARS SUB-GROUP
Number analyzed (Participants) | 160 | 136
Ratio | 45.0 [37.2 to 54.5] | 23.4 [19.1 to 28.7]

5. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/2009 Strain of Influenza Disease
Description: Titres are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/CAL/7/09. The reference seropositivity cut-off value was ≥ 1:10.
Time Frame: At Day 0, 21 and 42
Population: The ATP cohort for immunogenicity at Day 42 included all eligible subjects, for whom 2 (for D21 Groups)/1 (for M6 Groups) doses of study vaccine were administered and assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 (for D21 Groups)/42 (for M6 Groups) days after second/first vaccine dose.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- GSK2340272A 18-60 Years (D21) GROUP: Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21 (D21).
- GSK2340272A > 60 Years (D21) GROUP: Healthy male or female adults, older than 60 years of age (>60), who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
- GSK2340272A 18-60 Years (M6) GROUP: Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Month 6 (M6).
- GSK2340272A > 60 Years (M6) GROUP: Healthy male or female adults, > 60 years of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Month 6 (M6).
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 87 | 83 | 67 | 48
Titers
  Flu A/CAL/7/2009, Day 0 | 8.9 [7.2 to 11.0] | 7.3 [6.3 to 8.5] | 9.3 [7.4 to 11.8] | 8.0 [6.6 to 9.8]
  Flu A/CAL/7/2009, Day 21 | 459.8 [374.2 to 565.1] | 168.2 [129.0 to 219.3] | 366.1 [266.7 to 502.7] | 187.5 [136.6 to 257.4]
  Flu A/CAL/7/2009, Day 42 | 771.8 [660.5 to 901.7] | 400.9 [329.3 to 488.2] | 297.6 [218.6 to 405.2] | 132.6 [94.3 to 186.6]

6. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/2009 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/CAL/7/09. The reference seropositivity cut-off value was ≥ 1:10.
Time Frame: At Day 182
Population: The ATP cohort for antibody persistence at Day 182 included all eligible subjects, who received at least 1 dose of study vaccine according to their treatment assignment, had not received a vaccine not specified or forbidden in the protocol and for whom assay results were available for the study vaccine antigen component at Month 6.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 85 | 83 | 56 | 30
Titers | 240.5 [193.6 to 298.8] | 97.8 [79.4 to 120.4] | 124.1 [88.1 to 174.8] | 48.6 [30.0 to 78.9]

7. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/2009 Strain of Influenza Disease
Description: as for outcome 6
Time Frame: At Day 203
Population: The ATP cohort for immunogenicity at Day 203 included all eligible subjects form the GSK2340272A M6 Groups, for whom 2 doses were administrated and for whom assay results were available for antibodies against H1N1 antigen for blood sample taken 21 days after the second dose at Day 182.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- GSK2340272A > 60 Years (M6) GROUP: GROUP Healthy male or female adults, > 60 years of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Month 6 (M6).
Arm/Group | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 48 | 28
Titers | 708.3 [546.2 to 918.5] | 512.1 [354.5 to 740.0]

8. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 6
Time Frame: At Day 364
Population: The ATP cohort for persistence at Day 364 included all evaluable subjects, who met all the eligibility criteria, complied with the procedures defined in the protocol during the entire study and with the intervals defined in the protocol for visit at Day 364. This cohort included subjects for whom assay results were available at Day 364.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 79 | 76 | 60 | 46
Titers | 107.8 [82.9 to 140.1] | 35.8 [28.0 to 45.7] | 155.5 [116.8 to 207.0] | 68.8 [51.2 to 92.5]

9. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies
Description: as for outcome 1
Time Frame: At Day 21 and 42
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 87 | 83 | 67 | 48
Participants
  Flu A/CAL/7/2009, Day 21 | 87 | 74 | 62 | 43
  Flu A/CAL/7/2009, Day 42 | 86 | 82 | 61 | 39

10. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies
Description: as for outcome 1
Time Frame: At Day 182
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 85 | 83 | 56 | 30
Participants | 79 | 72 | 47 | 17

11. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies
Description: as for outcome 1
Time Frame: At Day 203
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 48 | 28
Participants | 48 | 28

12. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies
Description: as for outcome 1
Time Frame: At Day 364
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 79 | 76 | 60 | 46
Participants | 60 | 31 | 54 | 34

13. Secondary Outcome: Number of Subjects Who Were Seroprotected (SPR) for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 2
Time Frame: At Days 0, 21 and 42
Population: The ATP cohort for immunogenicity at Day 42 included all eligible subjects, for whom 2 (for D21 Groups)/1 (for M6 Groups) doses of study vaccine was administered and assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 (for D21 Groups)/42 (for M6 Groups) days after second/first vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 87 | 83 | 67 | 48
Participants
  Flu A/California/7/2009, Day 0 | 11 | 6 | 10 | 1
  Flu A/California/7/2009, Day 21 | 87 | 75 | 63 | 46
  Flu A/California/7/2009, Day 42 | 87 | 83 | 64 | 43

14. Secondary Outcome: Number of Subjects Who Were Seroprotected (SPR) for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 2
Time Frame: At Day 182
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 85 | 83 | 56 | 30
Participants | 83 | 75 | 48 | 19

15. Secondary Outcome: Number of Subjects Who Were Seroprotected (SPR) for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 2
Time Frame: At Day 203
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 48 | 28
Participants | 48 | 28

16. Secondary Outcome: Number of Subjects Who Were Seroprotected (SPR) for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titre greater than or equal to (≥) 1:40, that usually is accepted as indicating protection. The CHMP criterion was fulfilled if the post-vaccination point estimate for SPR was > 70% in subjects 18 to 60 of age or > 60% for subjects above 60 years of age.
Time Frame: At Day 364
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 79 | 76 | 60 | 46
Participants | 65 | 38 | 56 | 37

17. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 4
Time Frame: At Day 21 and 42
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 87 | 83 | 67 | 48
Ratio
  Flu A/CAL/7/09, Day 21 | 51.6 [40.7 to 65.5] | 23.0 [17.7 to 29.9] | 39.2 [28.3 to 54.2] | 23.3 [16.6 to 32.7]
  Flu A/CAL/7/09, Day 42 | 86.7 [68.6 to 109.5] | 54.9 [43.4 to 69.3] | 31.9 [23.4 to 43.4] | 16.5 [11.8 to 23.0]

18. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 4
Time Frame: At Day 182
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 85 | 83 | 56 | 30
Ratio | 26.6 [20.8 to 34.0] | 13.4 [10.9 to 16.5] | 14.6 [10.8 to 19.7] | 6.1 [3.9 to 9.4]

19. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 4
Time Frame: At Day 203
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 48 | 28
Ratio | 79.0 [58.0 to 107.7] | 65.7 [41.4 to 104.1]

20. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 4
Time Frame: At Day 364
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 79 | 76 | 60 | 46
Ratio | 11.9 [9.2 to 15.5] | 4.8 [3.8 to 6.1] | 17.3 [13.0 to 23.0] | 8.3 [6.0 to 11.3]

21. Secondary Outcome: Titers for Serum Neutralizing Antibodies Against Flu A/Netherlands/602/09 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/Neth/602/09. The reference seropositivity cut-off value was ≥ 1:8.
Time Frame: At Days 0, 21 and 42
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 24 | 24 | 19 | 18
Titers
  Flu A/Netherlands/602/09, Day 0 | 6.0 [4.2 to 8.6] | 10.2 [7.0 to 14.8] | 5.5 [4.1 to 7.4] | 17.9 [11.3 to 28.5]
  Flu A/Netherlands/602/09, Day 21 | 163.0 [84.3 to 315.2] | 96.4 [56.0 to 166.1] | 164.2 [64.0 to 420.7] | 168.3 [86.3 to 328.3]
  Flu A/Netherlands/602/09, Day 42 | 408.2 [257.0 to 648.4] | 207.8 [136.0 to 317.4] | 165.3 [70.7 to 386.1] | 105.0 [58.3 to 189.3]

22. Secondary Outcome: Percentage of Seroconverted Subjects for Serum Neutralizing Antibodies Against Flu A/Netherlands/602/09
Description: Seroconversion was defined as: For initially seronegative subjects, antibody titer ≥ 1:40 after vaccination; For initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was Flu A/Netherlands/602/09. The Committee for Medicinal Products for Human Use (CHMP) criterion was fulfilled if the point estimate for SCR was > 40% in subjects 18 to 60 years of age or > 30% for subjects above 60 years of age.
Time Frame: At Day 21 and 42
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 24 | 24 | 19 | 18
Percentage of subjects
  Flu A/Netherlands/602/09, Day 21 | 75.0 [53.3 to 90.2] | 62.5 [40.6 to 81.2] | 84.2 [60.4 to 96.6] | 61.1 [35.7 to 82.7]
  Flu A/Netherlands/602/09, Day 42 | 100 [85.8 to 100] | 87.5 [67.6 to 97.3] | 84.2 [60.4 to 96.6] | 61.1 [35.7 to 82.7]

23. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = significant pain at rest; prevented normal activities as assessed by inability to attend/do work or school. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following first dose - Interim Analysis posted at Day 42
Population: The Total Vaccinated cohort (TVc) included all subjects with at least 1 vaccine administration documented, who filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 YEARS SUB-GROUP | GSK2340272A > 60 YEARS SUB-GROUP
Number analyzed (Participants) | 162 | 142
Participants
  Any Pain | 154 | 106
  Grade 3 Pain | 0 | 2
  Any Redness | 18 | 9
  Grade 3 Redness | 0 | 0
  Any Swelling | 17 | 7
  Grade 3 Swelling | 0 | 0

24. Secondary Outcome: Duration of Solicited Local Symptoms Occurring in Response to Individual Doses
Description: The number of days with any solicited local symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following first dose - Interim Analysis posted at Day 42
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses
Arm/Group | GSK2340272A 18-60 YEARS SUB-GROUP | GSK2340272A > 60 YEARS SUB-GROUP
Number analyzed (Participants) | 162 | 142
Number analyzed (Doses) | 154 | 106
Days
  Pain | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
  Redness: number analyzed (Doses) | 18 | 9
  Redness | 2.0 [2.0 to 4.0] | 2.0 [2.0 to 3.0]
  Swelling: number analyzed (Doses) | 17 | 7
  Swelling | 3.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]

25. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: as for outcome 23
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses - Interim Analysis posted at Day 42
Population: The Total Vaccinated cohort (TVc) included all subjects from the GSK2340272A D21 Groups with at least 1 vaccine administration documented, who filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 YEARS (D21) GROUP | GSK2340272A > 60 YEARS (D21) GROUP
Number analyzed (Participants) | 92 | 90
Participants
  Any Pain, Dose 1 | 87 | 71
  Grade 3 Pain, Dose 1 | 0 | 2
  Any Redness, Dose 1 | 10 | 8
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 11 | 6
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 90 | 84
  Any Pain, Dose 2 | 80 | 62
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 90 | 84
  Grade 3 Pain, Dose 2 | 2 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 90 | 84
  Any Redness, Dose 2 | 6 | 11
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 90 | 84
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 90 | 84
  Any Swelling, Dose 2 | 8 | 10
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 90 | 84
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Across doses | 91 | 78
  Grade 3 Pain, Across doses | 2 | 2
  Any Redness, Across doses | 14 | 17
  Grade 3 Redness, Across doses | 0 | 0
  Any Swelling, Across doses | 15 | 15
  Grade 3 Swelling, Across doses | 0 | 0

26. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: as for outcome 23
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 92 | 90 | 70 | 52
Participants
  Any Pain, Dose 1 | 87 | 71 | 67 | 35
  Grade 3 Pain, Dose 1 | 0 | 2 | 0 | 0
  Any Redness, Dose 1 | 10 | 8 | 8 | 1
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 0
  Any Swelling, Dose 1 | 11 | 6 | 6 | 1
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 45
  Any Pain, Dose 2 | 80 | 62 | 54 | 26
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 45
  Grade 3 Pain, Dose 2 | 2 | 0 | 3 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 45
  Any Redness, Dose 2 | 6 | 11 | 6 | 3
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 45
  Grade 3 Redness, Dose 2 | 0 | 0 | 2 | 1
  Any Swelling, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 45
  Any Swelling, Dose 2 | 8 | 10 | 10 | 4
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 45
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 0
  Any Pain, Across doses | 91 | 78 | 68 | 40
  Grade 3 Pain, Across doses | 2 | 2 | 3 | 0
  Any Redness, Across doses | 14 | 17 | 13 | 4
  Grade 3 Redness, Across doses | 0 | 0 | 2 | 1
  Any Swelling, Across doses | 15 | 15 | 13 | 4
  Grade 3 Swelling, Across doses | 0 | 0 | 0 | 0

27. Secondary Outcome: Duration of Solicited Local Symptoms Occurring in Response to Individual Doses
Description: The number of days with any solicited local symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 92 | 90 | 70 | 52
Number analyzed (Doses) | 87 | 71 | 67 | 35
Days
  Pain, post-Dose 1 | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [1.0 to 4.0]
  Pain, post-Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 45
  Pain, post-Dose 2: number analyzed (Doses) | 80 | 62 | 54 | 26
  Pain, post-Dose 2 | 3.0 [2.0 to 3.5] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 3.0]
  Redness, post-Dose 1: number analyzed (Doses) | 10 | 8 | 8 | 1
  Redness, post-Dose 1 | 2.5 [1.0 to 4.0] | 2.0 [1.5 to 3.5] | 2.0 [2.0 to 3.5] | 3.0 [3.0 to 3.0]
  Redness, post-Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 45
  Redness, post-Dose 2: number analyzed (Doses) | 6 | 11 | 6 | 3
  Redness, post-Dose 2 | 2.5 [1.0 to 3.0] | 1.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 4.0 [3.0 to 6.0]
  Swelling, post-Dose 1: number analyzed (Doses) | 11 | 6 | 6 | 1
  Swelling, post-Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 3.0] | 3.0 [3.0 to 4.0] | 6.0 [6.0 to 6.0]
  Swelling, post-Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 45
  Swelling, post-Dose 2: number analyzed (Doses) | 8 | 10 | 10 | 4
  Swelling, post-Dose 2 | 2.0 [1.0 to 3.0] | 3.0 [1.0 to 4.0] | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 4.5]

28. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were Fatigue, Headache, Joint pain at other location, Muscle aches, Shivering, Sweating and Fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = general symptom that prevented normal everyday activities as assessed by inability to attend/do work or school, or required intervention of a physician/healthcare provider. Grade 3 fever = temperature ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following first dose - Interim Analysis posted at Day 42
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 YEARS SUB-GROUP | GSK2340272A > 60 YEARS SUB-GROUP
Number analyzed (Participants) | 162 | 142
Participants
  Any Fatigue | 67 | 44
  Grade 3 Fatigue | 1 | 0
  Related Fatigue | 56 | 34
  Any Headache | 56 | 29
  Grade 3 Headache | 1 | 1
  Related Headache | 43 | 23
  Any Joint pain | 31 | 27
  Grade 3 Joint pain | 0 | 0
  Related Joint pain | 26 | 20
  Any Muscle aches | 66 | 41
  Grade 3 Muscle aches | 0 | 1
  Related Muscle aches | 56 | 35
  Any Shivering | 31 | 18
  Grade 3 Shivering | 0 | 1
  Related Shivering | 22 | 11
  Any Sweating | 19 | 17
  Grade 3 Sweating | 1 | 0
  Related Sweating | 13 | 9
  Any Temperature | 3 | 2
  Grade 3 Temperature | 0 | 0
  Related Temperature | 1 | 0

29. Secondary Outcome: Duration of Solicited General Symptoms Occurring in Response to Individual Doses
Description: The number of days with any solicited general symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following first dose - Interim analysis posted at Day 42
Population: The Total Vaccinated cohort (TVc) included all subjects with at least 1 vaccine administrated documented, who filled in their symptom sheets.
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses
Arm/Group | GSK2340272A 18-60 YEARS SUB-GROUP | GSK2340272A > 60 YEARS SUB-GROUP
Number analyzed (Participants) | 162 | 142
Number analyzed (Doses) | 67 | 44
Days
  Fatigue | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Headache: number analyzed (Doses) | 56 | 29
  Headache | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0]
  Joint pain: number analyzed (Doses) | 31 | 27
  Joint pain | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Muscle aches: number analyzed (Doses) | 66 | 41
  Muscle aches | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Sweating: number analyzed (Doses) | 19 | 17
  Sweating | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Shivering: number analyzed (Doses) | 31 | 18
  Shivering | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Temperature: number analyzed (Doses) | 3 | 3
  Temperature | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]

30. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were Fatigue, Headache, Joint pain at other location, Muscle aches, Shivering, Sweating and Fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade or their relationship to vaccination. Grade 3 symptom = general symptom that prevented normal everyday activities as assessed by inability to attend/do work or school, or required intervention of a physician/healthcare provider. Grade 3 fever = temperature ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: as for outcome 25
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP
Number analyzed (Participants) | 92 | 90
Participants
  Any Fatigue, Dose 1 | 40 | 26
  Grade 3 Fatigue, Dose 1 | 0 | 0
  Related Fatigue, Dose 1 | 35 | 22
  Any Headache, Dose 1 | 34 | 20
  Grade 3 Headache, Dose 1 | 0 | 1
  Related Headache, Dose 1 | 30 | 17
  Any Joint pain, Dose 1 | 21 | 19
  Grade 3 Joint pain, Dose 1 | 0 | 0
  Related Joint pain, Dose 1 | 17 | 15
  Any Muscle aches, Dose 1 | 43 | 26
  Grade 3 Muscle aches, Dose 1 | 0 | 0
  Related Muscle aches, Dose 1 | 36 | 23
  Any Shivering, Dose 1 | 17 | 12
  Grade 3 Shivering, Dose 1 | 0 | 1
  Related Shivering, Dose 1 | 13 | 8
  Any Sweating, Dose 1 | 12 | 10
  Grade 3 Sweating, Dose 1 | 1 | 0
  Related Sweating, Dose 1 | 9 | 6
  Any Temperature, Dose 1 | 1 | 1
  Grade 3 Temperature, Dose 1 | 0 | 0
  Related Temperature, Dose 1 | 0 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 90 | 84
  Any Fatigue, Dose 2 | 48 | 27
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 90 | 84
  Grade 3 Fatigue, Dose 2 | 3 | 1
  Related Fatigue, Dose 2: number analyzed (Participants) | 90 | 84
  Related Fatigue, Dose 2 | 41 | 18
  Any Headache, Dose 2: number analyzed (Participants) | 90 | 84
  Any Headache, Dose 2 | 41 | 19
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 90 | 84
  Grade 3 Headache, Dose 2 | 1 | 1
  Related Headache, Dose 2: number analyzed (Participants) | 90 | 84
  Related Headache, Dose 2 | 36 | 12
  Any Joint pain, Dose 2: number analyzed (Participants) | 90 | 84
  Any Joint pain, Dose 2 | 17 | 21
  Grade 3 Joint pain, Dose 2: number analyzed (Participants) | 90 | 84
  Grade 3 Joint pain, Dose 2 | 0 | 0
  Related Joint pain, Dose 2: number analyzed (Participants) | 90 | 84
  Related Joint pain, Dose 2 | 13 | 17
  Any Muscle aches, Dose 2: number analyzed (Participants) | 90 | 84
  Any Muscle aches, Dose 2 | 38 | 25
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 90 | 84
  Grade 3 Muscle aches, Dose 2 | 0 | 0
  Related Muscle aches, Dose 2: number analyzed (Participants) | 90 | 84
  Related Muscle aches, Dose 2 | 31 | 19
  Any Shivering, Dose 2: number analyzed (Participants) | 90 | 84
  Any Shivering, Dose 2 | 26 | 13
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 90 | 84
  Grade 3 Shivering, Dose 2 | 1 | 1
  Related Shivering, Dose 2: number analyzed (Participants) | 90 | 84
  Related Shivering, Dose 2 | 24 | 9
  Any Sweating, Dose 2: number analyzed (Participants) | 90 | 84
  Any Sweating, Dose 2 | 19 | 13
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 90 | 84
  Grade 3 Sweating, Dose 2 | 1 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 90 | 84
  Related Sweating, Dose 2 | 17 | 8
  Any Temperature, Dose 2: number analyzed (Participants) | 90 | 84
  Any Temperature, Dose 2 | 6 | 5
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 90 | 84
  Grade 3 Temperature, Dose 2 | 0 | 2
  Related Temperature, Dose 2: number analyzed (Participants) | 90 | 84
  Related Temperature, Dose 2 | 5 | 4
  Any Fatigue, Across doses | 59 | 39
  Grade 3 Fatigue, Across doses | 3 | 1
  Related Fatigue, Across doses | 53 | 30
  Any Headache, Across doses | 53 | 30
  Grade 3 Headache, Across doses | 1 | 2
  Related Headache, Across doses | 46 | 23
  Any Joint pain, Across doses | 26 | 27
  Grade 3 Joint pain, Across doses | 0 | 0
  Related Joint pain, Across doses | 21 | 22
  Any Muscle aches, Across doses | 53 | 34
  Grade 3 Muscle aches, Across doses | 0 | 0
  Related Muscle aches, Across doses | 46 | 29
  Any Shivering, Across doses | 34 | 22
  Grade 3 Shivering, Across doses | 1 | 2
  Related Shivering, Across doses | 29 | 15
  Any Sweating, Across doses | 24 | 19
  Grade 3 Sweating, Across doses | 2 | 0
  Related Sweating, Across doses | 19 | 13
  Any Temperature, Across doses | 7 | 5
  Grade 3 Temperature, Across doses | 0 | 2
  Related Temperature, Across doses | 5 | 4

31. Secondary Outcome: Duration of Solicited General Symptoms Occurring in Response to Individual Doses
Description: The number of days with any solicited general symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses - Interim analysis posed at Day 42
Population: as for outcome 25
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP
Number analyzed (Participants) | 92 | 90
Number analyzed (Doses) | 88 | 53
Days
  Fatigue, post-Dose 1: number analyzed (Doses) | 40 | 26
  Fatigue, post-Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Fatigue, post-Dose 2: number analyzed (Participants) | 90 | 84
  Fatigue, post-Dose 2: number analyzed (Doses) | 48 | 27
  Fatigue, post-Dose 2 | 2.0 [1.0 to 2.5] | 2.0 [1.0 to 4.0]
  Fatigue, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Headache, post-Dose 1: number analyzed (Doses) | 34 | 20
  Headache, post-Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.5]
  Headache, post-Dose 2: number analyzed (Participants) | 90 | 84
  Headache, post-Dose 2: number analyzed (Doses) | 41 | 19
  Headache, post-Dose 2 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Headache, Overall/dose: number analyzed (Doses) | 75 | 39
  Headache, Overall/dose | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Joint pain, post-Dose 1: number analyzed (Doses) | 21 | 19
  Joint pain, post-Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Joint pain, post-Dose 2: number analyzed (Participants) | 90 | 84
  Joint pain, post-Dose 2: number analyzed (Doses) | 17 | 21
  Joint pain, post-Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Joint pain, Overall/dose: number analyzed (Doses) | 38 | 40
  Joint pain, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.5]
  Muscle aches, post-Dose 1: number analyzed (Doses) | 43 | 26
  Muscle aches, post-Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Muscle aches, post-Dose 2: number analyzed (Participants) | 90 | 84
  Muscle aches, post-Dose 2: number analyzed (Doses) | 38 | 25
  Muscle aches, post-Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 3.0]
  Muscle aches, Overall/dose: number analyzed (Doses) | 81 | 51
  Muscle aches, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Sweating, post-Dose 1: number analyzed (Doses) | 12 | 10
  Sweating, post-Dose 1 | 1.5 [1.0 to 2.5] | 2.0 [1.0 to 2.0]
  Sweating, post-Dose 2: number analyzed (Participants) | 90 | 84
  Sweating, post-Dose 2: number analyzed (Doses) | 19 | 13
  Sweating, post-Dose 2 | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Sweating, Overall/dose: number analyzed (Doses) | 31 | 23
  Sweating, Overall/dose | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Shivering, post-Dose 1: number analyzed (Doses) | 17 | 12
  Shivering, post-Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.5]
  Shivering, post-Dose 2: number analyzed (Participants) | 90 | 84
  Shivering, post-Dose 2: number analyzed (Doses) | 26 | 13
  Shivering, post-Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Shivering, Overall/dose: number analyzed (Doses) | 43 | 25
  Shivering, Overall/dose | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Temperature, post-Dose 1: number analyzed (Doses) | 1 | 1
  Temperature, post-Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Temperature, post-Dose 2: number analyzed (Participants) | 90 | 84
  Temperature, post-Dose 2: number analyzed (Doses) | 6 | 5
  Temperature, post-Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Temperature, Overall/dose: number analyzed (Doses) | 7 | 6
  Temperature, Overall/dose | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]

32. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were Fatigue, Headache, Joint pain at other location, Muscle aches, Shivering, Sweating and Fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = general symptom that prevented normal everyday activities as assessed by inability to attend/do work or school, or required intervention of a physician/healthcare provider. Grade 3 fever = temperature > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 92 | 90 | 70 | 52
Participants
  Any Fatigue, Dose 1 | 40 | 26 | 27 | 18
  Grade 3 Fatigue, Dose 1 | 0 | 0 | 1 | 0
  Related Fatigue, Dose 1 | 35 | 22 | 21 | 11
  Any Headache, Dose 1 | 34 | 20 | 22 | 9
  Grade 3 Headache, Dose 1 | 0 | 1 | 1 | 0
  Related Headache, Dose 1 | 29 | 17 | 13 | 6
  Any Joint pain, Dose 1 | 21 | 19 | 10 | 8
  Grade 3 Joint pain, Dose 1 | 0 | 0 | 0 | 0
  Related Joint pain, Dose 1 | 17 | 15 | 9 | 5
  Any Muscle aches, Dose 1 | 43 | 26 | 23 | 15
  Grade 3 Muscle aches, Dose 1 | 0 | 0 | 0 | 1
  Related Muscle aches, Dose 1 | 36 | 23 | 20 | 12
  Any Shivering, Dose 1 | 17 | 12 | 14 | 6
  Grade 3 Shivering, Dose 1 | 0 | 1 | 0 | 0
  Related Shivering, Dose 1 | 12 | 8 | 9 | 2
  Any Sweating, Dose 1 | 12 | 10 | 7 | 7
  Grade 3 Sweating, Dose 1 | 1 | 0 | 0 | 0
  Related Sweating, Dose 1 | 8 | 6 | 4 | 3
  Any Temperature, Dose 1 | 1 | 1 | 2 | 1
  Grade 3 Temperature, Dose 1 | 0 | 0 | 0 | 0
  Related Temperature, Dose 1 | 0 | 0 | 1 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Any Fatigue, Dose 2 | 49 | 27 | 31 | 13
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Grade 3 Fatigue, Dose 2 | 3 | 1 | 2 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Related Fatigue, Dose 2 | 42 | 18 | 31 | 11
  Any Headache, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Any Headache, Dose 2 | 41 | 19 | 21 | 11
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Grade 3 Headache, Dose 2 | 1 | 1 | 3 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Related Headache, Dose 2 | 36 | 12 | 19 | 9
  Any Joint pain, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Any Joint pain, Dose 2 | 18 | 21 | 16 | 12
  Grade 3 Joint pain, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Grade 3 Joint pain, Dose 2 | 0 | 0 | 0 | 0
  Related Joint pain, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Related Joint pain, Dose 2 | 14 | 17 | 16 | 7
  Any Muscle aches, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Any Muscle aches, Dose 2 | 39 | 25 | 31 | 15
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Grade 3 Muscle aches, Dose 2 | 0 | 0 | 1 | 0
  Related Muscle aches, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Related Muscle aches, Dose 2 | 32 | 19 | 28 | 10
  Any Shivering, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Any Shivering, Dose 2 | 26 | 13 | 11 | 7
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Grade 3 Shivering, Dose 2 | 1 | 1 | 0 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Related Shivering, Dose 2 | 24 | 9 | 11 | 4
  Any Sweating, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Any Sweating, Dose 2 | 19 | 14 | 8 | 4
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Grade 3 Sweating, Dose 2 | 1 | 0 | 0 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Related Sweating, Dose 2 | 17 | 9 | 8 | 2
  Any Temperature, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Any Temperature, Dose 2 | 6 | 5 | 1 | 0
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Grade 3 Temperature, Dose 2 | 0 | 2 | 0 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Related Temperature, Dose 2 | 5 | 4 | 1 | 0
  Any Fatigue, Across doses | 59 | 39 | 41 | 25
  Grade 3 Fatigue, Across doses | 3 | 1 | 3 | 0
  Related Fatigue, Across doses | 52 | 29 | 38 | 18
  Any Headache, Across doses | 53 | 30 | 31 | 15
  Grade 3 Headache, Across doses | 1 | 2 | 3 | 0
  Related Headache, Across doses | 45 | 22 | 24 | 12
  Any Joint pain, Across doses | 27 | 27 | 20 | 17
  Grade 3 Joint pain, Across doses | 0 | 0 | 0 | 0
  Related Joint pain, Across doses | 22 | 21 | 20 | 11
  Any Muscle aches, Across doses | 53 | 34 | 40 | 25
  Grade 3 Muscle aches, Across doses | 0 | 0 | 1 | 1
  Related Muscle aches, Across doses | 46 | 28 | 37 | 20
  Any Shivering, Across doses | 34 | 22 | 20 | 10
  Grade 3 Shivering, Across doses | 1 | 2 | 0 | 0
  Related Shivering, Across doses | 28 | 15 | 18 | 6
  Any Sweating, Across doses | 24 | 19 | 13 | 11
  Grade 3 Sweating, Across doses | 2 | 0 | 0 | 0
  Related Sweating, Across doses | 18 | 13 | 10 | 5
  Any Temperature, Across doses | 7 | 5 | 3 | 1
  Grade 3 Temperature, Across doses | 0 | 2 | 0 | 0
  Related Temperature, Across doses | 5 | 4 | 2 | 0

33. Secondary Outcome: Duration of Solicited General Symptoms Occurring in Response to Individual Doses
Description: The number of days with any solicited general symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 92 | 90 | 70 | 52
Number analyzed (Doses) | 49 | 27 | 31 | 18
Days
  Fatigue, post-Dose 1: number analyzed (Doses) | 40 | 26 | 27 | 18
  Fatigue, post-Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 1.5 [1.0 to 3.0]
  Fatigue, post-Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Fatigue, post-Dose 2: number analyzed (Doses) | 49 | 27 | 31 | 13
  Fatigue, post-Dose 2 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Headache, post-Dose 1: number analyzed (Doses) | 34 | 20 | 22 | 9
  Headache, post-Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.5] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0]
  Headache, post-Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Headache, post-Dose 2: number analyzed (Doses) | 41 | 19 | 21 | 11
  Headache, post-Dose 2 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 3.0 [1.0 to 4.0]
  Joint pain, post-Dose 1: number analyzed (Doses) | 21 | 19 | 10 | 8
  Joint pain, post-Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 3.0 [1.5 to 4.5]
  Joint pain, post-Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Joint pain, post-Dose 2: number analyzed (Doses) | 18 | 21 | 16 | 12
  Joint pain, post-Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0]
  Muscle aches, post-Dose 1: number analyzed (Doses) | 43 | 26 | 23 | 15
  Muscle aches, post-Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 4.0] | 2.0 [1.0 to 3.0]
  Muscle aches, post-Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Muscle aches, post-Dose 2: number analyzed (Doses) | 39 | 25 | 31 | 15
  Muscle aches, post-Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 3.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
  Sweating, post-Dose 1: number analyzed (Doses) | 12 | 10 | 7 | 7
  Sweating, post-Dose 1 | 1.5 [1.0 to 2.5] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Sweating, post-Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Sweating, post-Dose 2: number analyzed (Doses) | 19 | 14 | 8 | 4
  Sweating, post-Dose 2 | 2.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Shivering, post-Dose 1: number analyzed (Doses) | 17 | 12 | 14 | 6
  Shivering, post-Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.5] | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0]
  Shivering, post-Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Shivering, post-Dose 2: number analyzed (Doses) | 26 | 13 | 11 | 7
  Shivering, post-Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0]
  Temperature, post-Dose 1: number analyzed (Doses) | 1 | 1 | 2 | 1
  Temperature, post-Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Temperature, post-Dose 2: number analyzed (Participants) | 91 | 85 | 60 | 44
  Temperature, post-Dose 2: number analyzed (Doses) | 6 | 5 | 1 | 0
  Temperature, post-Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 2.0 [2.0 to 2.0] |

34. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESIs)/ Potential Immune-mediated Diseases (pIMDs)
Description: An AESI/pIMD was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: From Day 0 up to Day 42 - Interim analysis posted at Day 42
Population: The Total Vaccinated cohort (TVc) included all subjects with at least 1 vaccine administrated documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 93 | 91 | 70 | 52
Participants | 0 | 0 | 0 | 0

35. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESIs)/ Potential Immune-mediated Diseases (pIMDs)
Description: as for outcome 34
Time Frame: From Day 0 up to Day 203 - Interim analysis posted at Day 182/203
Population: The Total Vaccinated cohort (TVc) included all subjects with at least 1 vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 93 | 91 | 70 | 52
Participants | 0 | 0 | 0 | 0

36. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESIs)/ Potential Immune-mediated Diseases (pIMDs)
Description: as for outcome 34
Time Frame: From Day 0 up to Day 364
Population: The Total Vaccinated cohort (TVc) included all subjects with at least 1 vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 93 | 91 | 70 | 52
Participants
  Any AESI(s) | 1 | 0 | 1 | 0
  Related AESI(s) | 0 | 0 | 0 | 0

37. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESIs)
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: From Day 0 up to Day 364
Population: The Total Vaccinated cohort (TVc) included all subjects with at least 1 vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 93 | 91 | 70 | 52
Participants
  Any AESI(s) | 0 | 1 | 1 | 0
  Related AESI(s) | 0 | 1 | 0 | 0

38. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESIs)/ Potential Immune-mediated Diseases (pIMDs)
Description: as for outcome 34
Time Frame: From Day 0 up to Day 546
Population: The Total Vaccinated cohort (TVc) included all subjects from the GSK2340272A M6 Groups with at least 1 vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 70 | 52
Participants
  Any AESI(s) | 1 | 0
  Related AESI(s) | 0 | 0

39. Secondary Outcome: Number of Subjects With Normal/Abnormal Biochemical and Haematological Levels
Description: Among biochemical and haematological parameters assessed were alanine aminotransferase [ALAT], alkaline phosphatase [AP], aspartate aminotransferase [ASAT], bilirubin [BIL], creatinine [CRE], blood urea nitrogen [BUN]. Levels of haematological/biochemical parameters assessed with respect to normal laboratory values were - unknown, below, within and above in subjects aged 18-60 years and > 6 years old.
Time Frame: At Day 0 and 21 - Interim analysis posted at Day 42
Population: The Total Vaccinated cohort (TVc) included all subjects with at least 1 vaccine administration documented and with laboratory results available for the laboratory parameter assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 YEARS SUB-GROUP | GSK2340272A > 60 YEARS SUB-GROUP
Number analyzed (Participants) | 163 | 143
Participants
  ALAT, Day 0 - Unknown | 0 | 2
  ALAT, Day 0 - Below | 4 | 0
  ALAT, Day 0 - Within | 144 | 129
  ALAT, Day 0 - Above | 13 | 12
  ALAT, Day 21 - Unknown: number analyzed (Participants) | 161 | 140
  ALAT, Day 21 - Unknown | 1 | 0
  ALAT, Day 21 - Below: number analyzed (Participants) | 161 | 140
  ALAT, Day 21 - Below | 3 | 0
  ALAT, Day 21 - Within: number analyzed (Participants) | 161 | 140
  ALAT, Day 21 - Within | 143 | 123
  ALAT, Day 21 - Above: number analyzed (Participants) | 161 | 140
  ALAT, Day 21 - Above | 12 | 14
  AP, Day 0 - Unknown | 1 | 0
  AP, Day 0 - Below | 7 | 5
  AP, Day 0 - Within | 150 | 135
  AP, Day 0 - Above | 3 | 3
  AP, Day 21 - Unknown: number analyzed (Participants) | 161 | 140
  AP, Day 21 - Unknown | 0 | 0
  AP, Day 21 - Below: number analyzed (Participants) | 161 | 140
  AP, Day 21 - Below | 8 | 5
  AP, Day 21 - Within: number analyzed (Participants) | 161 | 140
  AP, Day 21 - Within | 149 | 128
  AP, Day 21 - Above: number analyzed (Participants) | 161 | 140
  AP, Day 21 - Above | 2 | 4
  ASAT, Day 0 - Unknown | 0 | 2
  ASAT, Day 0 - Below | 2 | 1
  ASAT, Day 0 - Within | 149 | 130
  ASAT, Day 0 - Above | 10 | 10
  ASAT, Day 21 - Unknown: number analyzed (Participants) | 161 | 140
  ASAT, Day 21 - Unknown | 1 | 1
  ASAT, Day 21 - Below: number analyzed (Participants) | 161 | 140
  ASAT, Day 21 - Below | 0 | 1
  ASAT, Day 21 - Within: number analyzed (Participants) | 161 | 140
  ASAT, Day 21 - Within | 147 | 125
  ASAT, Day 21 - Above: number analyzed (Participants) | 161 | 140
  ASAT, Day 21 - Above | 11 | 10
  BIL, Day 0 - Unknown | 1 | 2
  BIL, Day 0 - Below | 0 | 0
  BIL, Day 0 - Within | 153 | 137
  BIL, Day 0 - Above | 7 | 4
  BIL, Day 21 - Unknown: number analyzed (Participants) | 161 | 140
  BIL, Day 21 - Unknown | 1 | 0
  BIL, Day 21 - Below: number analyzed (Participants) | 161 | 140
  BIL, Day 21 - Below | 0 | 0
  BIL, Day 21 - Within: number analyzed (Participants) | 161 | 140
  BIL, Day 21 - Within | 151 | 132
  BIL, Day 21 - Above: number analyzed (Participants) | 161 | 140
  BIL, Day 21 - Above | 7 | 5
  CRE, Day 0 - Unknown | 0 | 0
  CRE, Day 0 - Below | 5 | 2
  CRE, Day 0 - Within | 149 | 120
  CRE, Day 0 - Above | 7 | 21
  CRE, Day 21 - Unknown: number analyzed (Participants) | 161 | 140
  CRE, Day 21 - Unknown | 0 | 0
  CRE, Day 21 - Below: number analyzed (Participants) | 161 | 140
  CRE, Day 21 - Below | 5 | 3
  CRE, Day 21 - Within: number analyzed (Participants) | 161 | 140
  CRE, Day 21 - Within | 146 | 119
  CRE, Day 21 - Above: number analyzed (Participants) | 161 | 140
  CRE, Day 21 - Above | 8 | 15
  BUN, Day 0 - Unknown | 2 | 1
  BUN, Day 0 - Below | 1 | 3
  BUN, Day 0 - Within | 153 | 110
  BUN, Day 0 - Above | 5 | 29
  BUN, Day 21 - Unknown: number analyzed (Participants) | 161 | 140
  BUN, Day 21 - Unknown | 0 | 0
  BUN, Day 21 - Below: number analyzed (Participants) | 161 | 140
  BUN, Day 21 - Below | 0 | 2
  BUN, Day 21 - Within: number analyzed (Participants) | 161 | 140
  BUN, Day 21 - Within | 152 | 102
  BUN, Day 21 - Above: number analyzed (Participants) | 161 | 140
  BUN, Day 21 - Above | 7 | 33

40. Secondary Outcome: Number of Subjects With Normal/Abnormal Biochemical and Haematological Levels
Description: Among biochemical and haematological parameters assessed were alanine aminotransferase [ALAT], alkaline phosphatase [AP], aspartate aminotransferase [ASAT], bilirubin [BIL], creatinine [CRE], blood urea nitrogen [BUN]. Levels of haematological/biochemical parameters assessed with respect to normal laboratory values were - unknown, bellow, within and above in subjects aged 18-60 years and > 6 years old.
Time Frame: At Days 0, 21 and 42 - Interim analysis posted at Day 42
Population: The Total Vaccinated cohort (TVc) included all subjects from the GSK2340272A D21 Groups with at least 1 vaccine administration documented and with laboratory results available for the laboratory parameter assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP
Number analyzed (Participants) | 93 | 91
Participants
  ALAT, Day 0 - Unknown | 0 | 2
  ALAT, Day 0 - Below | 4 | 0
  ALAT, Day 0 - Within | 83 | 83
  ALAT, Day 0 - Above | 4 | 6
  ALAT, Day 21 - Unknown: number analyzed (Participants) | 91 | 88
  ALAT, Day 21 - Unknown | 1 | 0
  ALAT, Day 21 - Below: number analyzed (Participants) | 91 | 88
  ALAT, Day 21 - Below | 3 | 0
  ALAT, Day 21 - Within: number analyzed (Participants) | 91 | 88
  ALAT, Day 21 - Within | 83 | 74
  ALAT, Day 21 - Above: number analyzed (Participants) | 91 | 88
  ALAT, Day 21 - Above | 3 | 11
  ALAT, Day 42 - Unknown: number analyzed (Participants) | 92 | 86
  ALAT, Day 42 - Unknown | 0 | 0
  ALAT, Day 42 - Below: number analyzed (Participants) | 92 | 86
  ALAT, Day 42 - Below | 3 | 0
  ALAT, Day 42 - Within: number analyzed (Participants) | 92 | 86
  ALAT, Day 42 - Within | 84 | 79
  ALAT, Day 42 - Above: number analyzed (Participants) | 92 | 86
  ALAT, Day 42 - Above | 5 | 6
  AP, Day 0 - Unknown | 1 | 0
  AP, Day 0 - Below | 3 | 22
  AP, Day 0 - Within | 85 | 86
  AP, Day 0 - Above | 2 | 3
  AP, Day 21 - Unknown: number analyzed (Participants) | 91 | 88
  AP, Day 21 - Unknown | 0 | 0
  AP, Day 21 - Below: number analyzed (Participants) | 91 | 88
  AP, Day 21 - Below | 3 | 2
  AP, Day 21 - Within: number analyzed (Participants) | 91 | 88
  AP, Day 21 - Within | 86 | 79
  AP, Day 21 - Above: number analyzed (Participants) | 91 | 88
  AP, Day 21 - Above | 1 | 4
  AP, Day 42 - Unknown: number analyzed (Participants) | 92 | 86
  AP, Day 42 - Unknown | 0 | 0
  AP, Day 42 - Below: number analyzed (Participants) | 92 | 86
  AP, Day 42 - Below | 2 | 2
  AP, Day 42 - Within: number analyzed (Participants) | 92 | 86
  AP, Day 42 - Within | 88 | 82
  AP, Day 42 - Above: number analyzed (Participants) | 92 | 86
  AP, Day 42 - Above | 2 | 1
  ASAT, Day 0 - Unknown | 0 | 2
  ASAT, Day 0 - Below | 1 | 1
  ASAT, Day 0 - Within | 87 | 81
  ASAT, Day 0 - Above | 3 | 7
  ASAT, Day 21 - Unknown: number analyzed (Participants) | 91 | 88
  ASAT, Day 21 - Unknown | 1 | 1
  ASAT, Day 21 - Below: number analyzed (Participants) | 91 | 88
  ASAT, Day 21 - Below | 0 | 1
  ASAT, Day 21 - Within: number analyzed (Participants) | 91 | 88
  ASAT, Day 21 - Within | 85 | 75
  ASAT, Day 21 - Above: number analyzed (Participants) | 91 | 88
  ASAT, Day 21 - Above | 4 | 8
  ASAT, Day 42 - Unknown: number analyzed (Participants) | 92 | 86
  ASAT, Day 42 - Unknown | 0 | 0
  ASAT, Day 42 - Below: number analyzed (Participants) | 92 | 86
  ASAT, Day 42 - Below | 0 | 0
  ASAT, Day 42 - Within: number analyzed (Participants) | 92 | 86
  ASAT, Day 42 - Within | 88 | 79
  ASAT, Day 42 - Above: number analyzed (Participants) | 92 | 86
  ASAT, Day 42 - Above | 4 | 6
  BIL, Day 0 - Unknown | 0 | 2
  BIL, Day 0 - Below | 0 | 0
  BIL, Day 0 - Within | 86 | 88
  BIL, Day 0 - Above | 5 | 1
  BIL, Day 21 - Unknown: number analyzed (Participants) | 91 | 88
  BIL, Day 21 - Unknown | 1 | 0
  BIL, Day 21 - Below: number analyzed (Participants) | 91 | 88
  BIL, Day 21 - Below | 0 | 0
  BIL, Day 21 - Within: number analyzed (Participants) | 91 | 88
  BIL, Day 21 - Within | 86 | 83
  BIL, Day 21 - Above: number analyzed (Participants) | 91 | 88
  BIL, Day 21 - Above | 3 | 2
  BIL, Day 42 - Unknown: number analyzed (Participants) | 92 | 86
  BIL, Day 42 - Unknown | 0 | 0
  BIL, Day 42 - Below: number analyzed (Participants) | 92 | 86
  BIL, Day 42 - Below | 0 | 0
  BIL, Day 42 - Within: number analyzed (Participants) | 92 | 86
  BIL, Day 42 - Within | 89 | 84
  BIL, Day 42 - Above: number analyzed (Participants) | 92 | 86
  BIL, Day 42 - Above | 3 | 1
  CRE, Day 0 - Unknown | 0 | 0
  CRE, Day 0 - Below | 1 | 1
  CRE, Day 0 - Within | 86 | 75
  CRE, Day 0 - Above | 4 | 15
  CRE, Day 21 - Unknown: number analyzed (Participants) | 91 | 88
  CRE, Day 21 - Unknown | 0 | 0
  CRE, Day 21 - Below: number analyzed (Participants) | 91 | 88
  CRE, Day 21 - Below | 2 | 0
  CRE, Day 21 - Within: number analyzed (Participants) | 91 | 88
  CRE, Day 21 - Within | 83 | 73
  CRE, Day 21 - Above: number analyzed (Participants) | 91 | 88
  CRE, Day 21 - Above | 5 | 12
  CRE, Day 42 - Unknown: number analyzed (Participants) | 92 | 86
  CRE, Day 42 - Unknown | 0 | 0
  CRE, Day 42 - Below: number analyzed (Participants) | 92 | 86
  CRE, Day 42 - Below | 5 | 2
  CRE, Day 42 - Within: number analyzed (Participants) | 92 | 86
  CRE, Day 42 - Within | 84 | 75
  CRE, Day 42 - Above: number analyzed (Participants) | 92 | 86
  CRE, Day 42 - Above | 3 | 8
  BUN, Day 0 - Unknown | 2 | 1
  BUN, Day 0 - Below | 1 | 1
  BUN, Day 0 - Within | 87 | 67
  BUN, Day 0 - Above | 1 | 22
  BUN, Day 21 - Unknown: number analyzed (Participants) | 91 | 88
  BUN, Day 21 - Unknown | 0 | 0
  BUN, Day 21 - Below: number analyzed (Participants) | 91 | 88
  BUN, Day 21 - Below | 0 | 1
  BUN, Day 21 - Within: number analyzed (Participants) | 91 | 88
  BUN, Day 21 - Within | 87 | 60
  BUN, Day 21 - Above: number analyzed (Participants) | 91 | 88
  BUN, Day 21 - Above | 3 | 24
  BUN, Day 42 - Unknown: number analyzed (Participants) | 92 | 86
  BUN, Day 42 - Unknown | 3 | 2
  BUN, Day 42 - Below: number analyzed (Participants) | 92 | 86
  BUN, Day 42 - Below | 0 | 0
  BUN, Day 42 - Within: number analyzed (Participants) | 92 | 86
  BUN, Day 42 - Within | 84 | 66
  BUN, Day 42 - Above: number analyzed (Participants) | 92 | 86
  BUN, Day 42 - Above | 5 | 17

41. Secondary Outcome: Number of Subjects With Normal/Abnormal Biochemical and Haematological Levels
Description: as for outcome 40
Time Frame: At Days 0, 21, 42 and 182
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 93 | 91 | 70 | 52
Participants
  ALAT, Day 0 - Unknown | 0 | 2 | 0 | 0
  ALAT, Day 0 - Below | 4 | 0 | 0 | 0
  ALAT, Day 0 - Within | 83 | 83 | 60 | 46
  ALAT, Day 0 - Above | 4 | 5 | 9 | 6
  ALAT, Day 21 - Unknown: number analyzed (Participants) | 91 | 88 | 70 | 52
  ALAT, Day 21 - Unknown | 1 | 0 | 0 | 0
  ALAT, Day 21 - Below: number analyzed (Participants) | 91 | 88 | 70 | 52
  ALAT, Day 21 - Below | 3 | 0 | 0 | 0
  ALAT, Day 21 - Within: number analyzed (Participants) | 91 | 88 | 70 | 52
  ALAT, Day 21 - Within | 83 | 74 | 59 | 49
  ALAT, Day 21 - Above: number analyzed (Participants) | 91 | 88 | 70 | 52
  ALAT, Day 21 - Above | 3 | 10 | 9 | 3
  ALAT, Day 42 - Unknown: number analyzed (Participants) | 92 | 86 | 68 | 52
  ALAT, Day 42 - Unknown | 0 | 0 | 0 | 0
  ALAT, Day 42 - Below: number analyzed (Participants) | 92 | 86 | 68 | 52
  ALAT, Day 42 - Below | 3 | 0 | 0 | 0
  ALAT, Day 42 - Within: number analyzed (Participants) | 92 | 86 | 68 | 52
  ALAT, Day 42 - Within | 84 | 79 | 61 | 47
  ALAT, Day 42 - Above: number analyzed (Participants) | 92 | 86 | 68 | 52
  ALAT, Day 42 - Above | 5 | 6 | 7 | 4
  ALAT, Day 182 - Unknown: number analyzed (Participants) | 88 | 85 | 63 | 47
  ALAT, Day 182 - Unknown | 0 | 0 | 0 | 0
  ALAT, Day 182 - Below: number analyzed (Participants) | 88 | 85 | 63 | 47
  ALAT, Day 182 - Below | 2 | 0 | 0 | 0
  ALAT, Day 182 - Within: number analyzed (Participants) | 88 | 85 | 63 | 47
  ALAT, Day 182 - Within | 84 | 76 | 53 | 42
  ALAT, Day 182 - Above: number analyzed (Participants) | 88 | 85 | 63 | 47
  ALAT, Day 182 - Above | 2 | 9 | 10 | 4
  AP, Day 0 - Unknown | 1 | 0 | 0 | 0
  AP, Day 0 - Below | 3 | 2 | 4 | 3
  AP, Day 0 - Within | 85 | 86 | 64 | 49
  AP, Day 0 - Above | 2 | 2 | 1 | 0
  AP, Day 21 - Unknown: number analyzed (Participants) | 91 | 88 | 70 | 52
  AP, Day 21 - Unknown | 0 | 0 | 0 | 0
  AP, Day 21 - Below: number analyzed (Participants) | 91 | 88 | 70 | 52
  AP, Day 21 - Below | 3 | 2 | 5 | 3
  AP, Day 21 - Within: number analyzed (Participants) | 91 | 88 | 70 | 52
  AP, Day 21 - Within | 86 | 79 | 62 | 49
  AP, Day 21 - Above: number analyzed (Participants) | 91 | 88 | 70 | 52
  AP, Day 21 - Above | 1 | 3 | 1 | 0
  AP, Day 42 - Unknown: number analyzed (Participants) | 92 | 86 | 68 | 52
  AP, Day 42 - Unknown | 0 | 0 | 1 | 0
  AP, Day 42 - Below: number analyzed (Participants) | 92 | 86 | 68 | 52
  AP, Day 42 - Below | 2 | 2 | 3 | 4
  AP, Day 42 - Within: number analyzed (Participants) | 92 | 86 | 68 | 52
  AP, Day 42 - Within | 88 | 82 | 63 | 47
  AP, Day 42 - Above: number analyzed (Participants) | 92 | 86 | 68 | 52
  AP, Day 42 - Above | 2 | 1 | 1 | 0
  AP, Day 182 - Unknown: number analyzed (Participants) | 88 | 85 | 63 | 47
  AP, Day 182 - Unknown | 1 | 1 | 0 | 1
  AP, Day 182 - Below: number analyzed (Participants) | 88 | 85 | 63 | 47
  AP, Day 182 - Below | 4 | 2 | 1 | 2
  AP, Day 182 - Within: number analyzed (Participants) | 88 | 85 | 63 | 47
  AP, Day 182 - Within | 81 | 81 | 62 | 43
  AP, Day 182 - Above: number analyzed (Participants) | 88 | 85 | 63 | 47
  AP, Day 182 - Above | 2 | 1 | 0 | 0
  ASAT, Day 0 - Unknown | 0 | 2 | 0 | 0
  ASAT, Day 0 - Below | 1 | 0 | 1 | 0
  ASAT, Day 0 - Within | 87 | 81 | 61 | 49
  ASAT, Day 0 - Above | 3 | 7 | 7 | 3
  ASAT, Day 21 - Unknown: number analyzed (Participants) | 91 | 88 | 70 | 52
  ASAT, Day 21 - Unknown | 1 | 1 | 0 | 0
  ASAT, Day 21 - Below: number analyzed (Participants) | 91 | 88 | 70 | 52
  ASAT, Day 21 - Below | 0 | 0 | 0 | 0
  ASAT, Day 21 - Within: number analyzed (Participants) | 91 | 88 | 70 | 52
  ASAT, Day 21 - Within | 85 | 75 | 61 | 50
  ASAT, Day 21 - Above: number analyzed (Participants) | 91 | 88 | 70 | 52
  ASAT, Day 21 - Above | 4 | 8 | 7 | 2
  ASAT, Day 42 - Unknown: number analyzed (Participants) | 92 | 86 | 68 | 52
  ASAT, Day 42 - Unknown | 0 | 0 | 0 | 0
  ASAT, Day 42 - Below: number analyzed (Participants) | 92 | 86 | 68 | 52
  ASAT, Day 42 - Below | 0 | 0 | 1 | 0
  ASAT, Day 42 - Within: number analyzed (Participants) | 92 | 86 | 68 | 52
  ASAT, Day 42 - Within | 88 | 79 | 58 | 49
  ASAT, Day 42 - Above: number analyzed (Participants) | 92 | 86 | 68 | 52
  ASAT, Day 42 - Above | 4 | 6 | 9 | 2
  ASAT, Day 182 - Unknown: number analyzed (Participants) | 88 | 85 | 63 | 47
  ASAT, Day 182 - Unknown | 0 | 0 | 0 | 0
  ASAT, Day 182 - Below: number analyzed (Participants) | 88 | 85 | 63 | 47
  ASAT, Day 182 - Below | 0 | 0 | 0 | 0
  ASAT, Day 182 - Within: number analyzed (Participants) | 88 | 85 | 63 | 47
  ASAT, Day 182 - Within | 86 | 79 | 59 | 44
  ASAT, Day 182 - Above: number analyzed (Participants) | 88 | 85 | 63 | 47
  ASAT, Day 182 - Above | 2 | 6 | 4 | 2
  BIL, Day 0 - Unknown | 0 | 2 | 1 | 0
  BIL, Day 0 - Below | 0 | 0 | 0 | 0
  BIL, Day 0 - Within | 86 | 87 | 66 | 49
  BIL, Day 0 - Above | 5 | 1 | 2 | 3
  BIL, Day 21 - Unknown: number analyzed (Participants) | 91 | 88 | 70 | 52
  BIL, Day 21 - Unknown | 1 | 0 | 0 | 0
  BIL, Day 21 - Below: number analyzed (Participants) | 91 | 88 | 70 | 52
  BIL, Day 21 - Below | 0 | 0 | 0 | 0
  BIL, Day 21 - Within: number analyzed (Participants) | 91 | 88 | 70 | 52
  BIL, Day 21 - Within | 86 | 82 | 64 | 49
  BIL, Day 21 - Above: number analyzed (Participants) | 91 | 88 | 70 | 52
  BIL, Day 21 - Above | 3 | 2 | 4 | 3
  BIL, Day 42 - Unknown: number analyzed (Participants) | 92 | 86 | 68 | 52
  BIL, Day 42 - Unknown | 0 | 0 | 1 | 0
  BIL, Day 42 - Below: number analyzed (Participants) | 92 | 86 | 68 | 52
  BIL, Day 42 - Below | 0 | 0 | 0 | 0
  BIL, Day 42 - Within: number analyzed (Participants) | 92 | 86 | 68 | 52
  BIL, Day 42 - Within | 89 | 84 | 63 | 49
  BIL, Day 42 - Above: number analyzed (Participants) | 92 | 86 | 68 | 52
  BIL, Day 42 - Above | 3 | 1 | 4 | 2
  BIL, Day 182 - Unknown: number analyzed (Participants) | 88 | 85 | 63 | 47
  BIL, Day 182 - Unknown | 1 | 4 | 1 | 1
  BIL, Day 182 - Below: number analyzed (Participants) | 88 | 85 | 63 | 47
  BIL, Day 182 - Below | 0 | 0 | 0 | 0
  BIL, Day 182 - Within: number analyzed (Participants) | 88 | 85 | 63 | 47
  BIL, Day 182 - Within | 84 | 80 | 59 | 41
  BIL, Day 182 - Above: number analyzed (Participants) | 88 | 85 | 63 | 47
  BIL, Day 182 - Above | 3 | 1 | 3 | 4
  CRE, Day 0 - Unknown | 0 | 0 | 0 | 0
  CRE, Day 0 - Below | 1 | 1 | 4 | 1
  CRE, Day 0 - Within | 86 | 75 | 63 | 45
  CRE, Day 0 - Above | 4 | 14 | 2 | 6
  CRE, Day 21 - Unknown: number analyzed (Participants) | 91 | 88 | 70 | 52
  CRE, Day 21 - Unknown | 0 | 0 | 0 | 0
  CRE, Day 21 - Below: number analyzed (Participants) | 91 | 88 | 70 | 52
  CRE, Day 21 - Below | 2 | 0 | 3 | 3
  CRE, Day 21 - Within: number analyzed (Participants) | 91 | 88 | 70 | 52
  CRE, Day 21 - Within | 83 | 73 | 62 | 46
  CRE, Day 21 - Above: number analyzed (Participants) | 91 | 88 | 70 | 52
  CRE, Day 21 - Above | 5 | 11 | 3 | 3
  CRE, Day 42 - Unknown: number analyzed (Participants) | 92 | 86 | 68 | 52
  CRE, Day 42 - Unknown | 0 | 0 | 0 | 0
  CRE, Day 42 - Below: number analyzed (Participants) | 92 | 86 | 68 | 52
  CRE, Day 42 - Below | 5 | 2 | 4 | 1
  CRE, Day 42 - Within: number analyzed (Participants) | 92 | 86 | 68 | 52
  CRE, Day 42 - Within | 84 | 75 | 62 | 47
  CRE, Day 42 - Above: number analyzed (Participants) | 92 | 86 | 68 | 52
  CRE, Day 42 - Above | 3 | 8 | 2 | 3
  CRE, Day 182 - Unknown: number analyzed (Participants) | 88 | 85 | 63 | 47
  CRE, Day 182 - Unknown | 0 | 0 | 0 | 0
  CRE, Day 182 - Below: number analyzed (Participants) | 88 | 85 | 63 | 47
  CRE, Day 182 - Below | 4 | 0 | 2 | 1
  CRE, Day 182 - Within: number analyzed (Participants) | 88 | 85 | 63 | 47
  CRE, Day 182 - Within | 81 | 76 | 57 | 42
  CRE, Day 182 - Above: number analyzed (Participants) | 88 | 85 | 63 | 47
  CRE, Day 182 - Above | 3 | 9 | 4 | 3
  BUN, Day 0 - Unknown | 2 | 1 | 0 | 0
  BUN, Day 0 - Below | 1 | 0 | 0 | 2
  BUN, Day 0 - Within | 87 | 67 | 65 | 43
  BUN, Day 0 - Above | 1 | 22 | 4 | 7
  BUN, Day 21 - Unknown: number analyzed (Participants) | 91 | 88 | 70 | 52
  BUN, Day 21 - Unknown | 0 | 0 | 0 | 0
  BUN, Day 21 - Below: number analyzed (Participants) | 91 | 88 | 70 | 52
  BUN, Day 21 - Below | 0 | 0 | 0 | 1
  BUN, Day 21 - Within: number analyzed (Participants) | 91 | 88 | 70 | 52
  BUN, Day 21 - Within | 87 | 60 | 64 | 42
  BUN, Day 21 - Above: number analyzed (Participants) | 91 | 88 | 70 | 52
  BUN, Day 21 - Above | 3 | 24 | 4 | 9
  BUN, Day 42 - Unknown: number analyzed (Participants) | 92 | 86 | 68 | 52
  BUN, Day 42 - Unknown | 3 | 2 | 2 | 1
  BUN, Day 42 - Below: number analyzed (Participants) | 92 | 86 | 68 | 52
  BUN, Day 42 - Below | 0 | 0 | 1 | 1
  BUN, Day 42 - Within: number analyzed (Participants) | 92 | 86 | 68 | 52
  BUN, Day 42 - Within | 84 | 66 | 60 | 43
  BUN, Day 42 - Above: number analyzed (Participants) | 92 | 86 | 68 | 52
  BUN, Day 42 - Above | 5 | 17 | 5 | 6
  BUN, Day 182 - Unknown: number analyzed (Participants) | 88 | 85 | 63 | 47
  BUN, Day 182 - Unknown | 1 | 2 | 1 | 1
  BUN, Day 182 - Below: number analyzed (Participants) | 88 | 85 | 63 | 47
  BUN, Day 182 - Below | 1 | 0 | 2 | 1
  BUN, Day 182 - Within: number analyzed (Participants) | 88 | 85 | 63 | 47
  BUN, Day 182 - Within | 81 | 59 | 54 | 36
  BUN, Day 182 - Above: number analyzed (Participants) | 88 | 85 | 63 | 47
  BUN, Day 182 - Above | 5 | 24 | 6 | 8

42. Secondary Outcome: Number of Subjects With Normal/Abnormal Biochemical and Haematological Levels
Description: as for outcome 40
Time Frame: At Day 364
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 85 | 83 | 62 | 47
Participants
  ALAT - Unknown | 0 | 1 | 0 | 0
  ALAT - Below | 2 | 0 | 0 | 0
  ALAT - Within | 79 | 77 | 57 | 45
  ALAT - Above | 4 | 5 | 5 | 2
  AP - Unknown | 0 | 0 | 0 | 0
  AP - Below | 3 | 0 | 0 | 2
  AP - Within | 82 | 82 | 62 | 45
  AP - Above | 0 | 1 | 0 | 0
  ASAT - Unknown | 0 | 0 | 0 | 0
  ASAT - Below | 1 | 0 | 5 | 0
  ASAT - Within | 81 | 77 | 55 | 46
  ASAT - Above | 3 | 6 | 2 | 1
  BIL - Unknown | 1 | 0 | 0 | 0
  BIL - Below | 0 | 0 | 0 | 0
  BIL - Within | 81 | 82 | 59 | 44
  BIL - Above | 3 | 1 | 3 | 3
  CRE - Unknown | 0 | 1 | 0 | 0
  CRE - Below | 2 | 0 | 4 | 2
  CRE - Within | 82 | 75 | 56 | 41
  CRE - Above | 1 | 7 | 2 | 4
  BUN - Unknown | 1 | 0 | 1 | 2
  BUN - Below | 0 | 0 | 2 | 1
  BUN - Within | 84 | 65 | 57 | 37
  BUN - Above | 0 | 18 | 2 | 7

43. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination. Note: GSK2340272A 18-60 years (D21) GROUP and GSK2340272A >60 years (D21) GROUP presents results after the 2 vaccine dose; GSK2340272A 18-60 years (M6) GROUP and GSK2340272A >60 years (M6) GROUP presents result after 1 vaccine dose.
Time Frame: Within the 42-day (Days 0-41) post vaccination period - Interim analysis posted at Day 42
Population: The Total Vaccinated cohort (TVc) included all subjects with at least 1 vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 93 | 91 | 70 | 52
Participants
  Any AE(s) | 40 | 38 | 27 | 11
  Grade 3 AE(s) | 6 | 6 | 6 | 1
  Related AE(s) | 11 | 15 | 5 | 2

44. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 21- days post-Dose 1 vaccination (Days 0-20 in both groups) and either 63 days post-Dose 2 vaccination (Days 21-84 in D21 groups) or 21 days post-Dose 2 vaccination (Day 182-203 in M6 groups) - Interim analysis at Day 182/203
Population: The Total Vaccinated cohort (TVc) included all subjects with at least 1 vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 93 | 91 | 70 | 52
Participants
  Any AE(s) | 52 | 53 | 30 | 15
  Grade 3 AE(s) | 10 | 9 | 6 | 2
  Related AE(s) | 12 | 15 | 10 | 5

45. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: as for outcome 44
Time Frame: Within the 21-days post-Dose 1 vaccination (Days 0-20 in both groups) and either 63 days post-Dose 2 vaccination (Days 21-84 in D21 groups) or 30 days post-Dose 2 vaccination (Days 182-212 in M6 groups)
Population: The Total Vaccinated cohort (TVc) included all subjects with at least 1 vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 93 | 91 | 70 | 52
Participants
  Any AE(s) | 52 | 53 | 35 | 16
  Grade 3 AE(s) | 10 | 9 | 6 | 2
  Related AE(s) | 12 | 15 | 13 | 5

46. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 up to Day 364
Population: The Total Vaccinated cohort (TVc) included all subjects with at least 1 vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (D21) GROUP | GSK2340272A > 60 Years (D21) GROUP | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 93 | 91 | 70 | 52
Participants | 4 | 7 | 4 | 2

47. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 46
Time Frame: From Day 0 up to Day 546
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 18-60 Years (M6) GROUP | GSK2340272A > 60 Years (M6) GROUP
Number analyzed (Participants) | 70 | 52
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: within the 21 days post-Dose 1 vaccination (Days 0-20 for all groups) and either 63 days post-Dose 2 vaccination (Days 21-84 for D21 groups) or 30 days post-Dose 2 vaccination (Days 182-212 for M6 groups); SAEs: during the entire study period (from Day 0 up to Day 364 for the D21 groups and up to Day 546 for M6 groups).
Arm/Group | GSK2340272A (D21) GROUP | GSK2340272A (M6) GROUP
All-Cause Mortality (participants affected / at risk) | 0/184 | 0/122
Serious Adverse Events (participants affected / at risk) | 11/184 | 8/122
Other Adverse Events (participants affected / at risk) | 174/184 | 117/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340272A (D21) GROUP (N=184) | GSK2340272A (M6) GROUP (N=122)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340272A (D21) GROUP (N=184) | GSK2340272A (M6) GROUP (N=122)
Arthralgia (Musculoskeletal and connective tissue disorders) | 55 (82) | 39 (51)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 8 (9)
Chills (General disorders) | 56 (68) | 32 (40)
Erythema (Skin and subcutaneous tissue disorders) | 31 (35) | 17 (18)
Fatigue (General disorders) | 99 (144) | 68 (92)
Headache (Nervous system disorders) | 88 (129) | 48 (77)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 43 (55) | 24 (26)
Myalgia (Musculoskeletal and connective tissue disorders) | 88 (134) | 65 (85)
Nasopharyngitis (Infections and infestations) | 20 (22) | 11 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7)
Pain (General disorders) | 169 (301) | 108 (183)
Pyrexia (General disorders) | 14 (15) | 7 (7)
Rhinitis (Infections and infestations) | 20 (22) | 9 (9)
Swelling (General disorders) | 30 (35) | 17 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.